CLINICAL TRIAL: NCT02264340
Title: EFFECTS OF EXERCISE AND RELAXATION TECHNIQUES ON TENSION-TYPE HEADACHE PAIN PARAMETERS OF UNIVERSITY STUDENTS; A RANDOMIZED AND CONTROLLED CLINICAL TRIAL
Brief Title: Effects of Exercise and Relaxation Techniques on Tension Headache Pain Parameters of University Students
Acronym: ERTTHU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Ángela Álvarez Melcón, Physiotherapist (Doctor), Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F(EFP)-003/2010
Record Dates: First submitted 2014-10-08; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Tension-Type Headache
Keywords: Tension-type headache; relaxation techniques; physiotherapy
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Relaxation technique
  Interventions: Behavioral: Relaxation technique Autogenic Training
- Experimental (Experimental): Combined treatment
  Interventions: Behavioral: Combined treatment Autogenic Training + Cervical exercises and postural correction

INTERVENTIONS:
Behavioral: Relaxation technique Autogenic Training — Autogenic Training
  Arms: Control
Behavioral: Combined treatment Autogenic Training + Cervical exercises and postural correction — Autogenic Training + Cervical exercises and postural correction
  Arms: Experimental

SUMMARY:
Tension headache is a common disabling disease and a worldwide public health problem. This research tries to demonstrate the efficacy of physical therapy, based on cervical training and postural self-correction instructions, which aims to increase the positive results obtained from traditional relaxation techniques (Schultz Autogenic Training). University students are selected, because headaches are very common in this sector of the population. The design is a non-pharmacological randomized controlled trial, with blinded evaluation of the response variables. The investigators compare two independent samples. One of them receives an only treatment (Autogenic Training) and the other group receives a combined program (Autogenic Training + specific cervical exercises and postural correction). Pain parameters (frequency, intensity and duration) and drug consumption are measured before treatment, and then, at 4 weeks and 3 months, to value the results.

ELIGIBILITY:
Inclusion Criteria:

* College students of Complutense University of Madrid, diagnosed with frequent episodic or chronic tension-type headache (according to the criteria of International Headache Society (IHS)).

Exclusion Criteria:

* Cases with other headaches
* Students with excessive state anxiety and / or trait anxiety (≥ 85 percentile, State-Trait Anxiety Inventory )
* Students that had received treatment for tension headache, based on physical exercise or relaxation techniques, in the last 6 months.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Frequency | 4 weeks
  Days with headache, during 4 weeks

SECONDARY OUTCOMES:
Intensity | 4 weeks
  Pain intensity (VAS: 1-10)
Duration | 4 weeks
  Hours a day with headache
Medication | 4 weeks
  Days in which person takes drugs for pain, during 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ángela Álvarez Melcón, Doctor, Principal Investigator — Universidad Complutense de Madrid